CLINICAL TRIAL: NCT01019811
Title: The Innervated Sensory Cross-finger Flap Based on the Dorsal Branch Artery for Reconstruction of Fingertip Degloving Injury
Brief Title: Innervated Sensory Cross-Finger Flap
Acronym: ISCF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Second Hospital of Tangshan (Other)
Responsible Party: Dequn Liu, The Second Hospital of Tangshan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STS-5xb-86
Record Dates: First submitted 2009-11-20; First posted 2009-11-25 (Estimated); Last update posted 2009-11-25 (Estimated); Status verified 2009-11

CONDITIONS: Transplantation
Keywords: Cross-finger flap; finger injuries; fingertip reconstruction; proper digital artery; proper digital nerve.
MeSH Terms: conditions — Finger Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: The innervated sensory cross-finger flap — The innervated sensory cross-finger flap is a modified method for repair fingertip degloving injury

SUMMARY:
The purpose of this study is to introduce a new operative technique for reconstruction of fingertip degloving injury.

DETAILED DESCRIPTION:
Incidence of fingertip degloving injury is common and can result in functional morbidity. A cross-finger flap based on the dorsal branch artery (DBA) including sensory nerve is a useful reconstructive technique.In our modification, the innervated sensory flap is vascularized by the DBA, both its pedicle is narrow and its coverage is extended, the projecting tip of exposed distal phalanx of adjacent digits therefore can be wrapped.

ELIGIBILITY:
Inclusion Criteria:

* the fingertip degloving injury including the thumb;
* age between 12 and 59 years;
* no life-threatening associated injuries.

Exclusion Criteria:

* age greater than 60 years;
* smoking;
* Dupuytren's contracture;
* peripheral arterial disease and other vascular disorders.

Ages: 12 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 16 (Actual)
Dates: Start 2001-05; Primary Completion 2006-05 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
static 2-point discrimination test and the range of motion are used for evaluation of outcomes | at least 4 months

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Hospital of Tangshan, Tangshan, Hebei, China

REFERENCES:
- [Derived] Zhang W, Zhang X, Liu Y, Xu T, Zhuang Y, Chen C. Repair of Fingertip Degloving Injuries Using the Extended Reverse Second Dorsal Metacarpal Artery Flap. Plast Reconstr Surg. 2024 Jul 1;154(1):133-141. doi: 10.1097/PRS.0000000000010939. Epub 2023 Jul 25. PMID 37498313